CLINICAL TRIAL: NCT00107679
Title: Anal Dysplasia: A Substudy of a Large, Simple Trial Comparing Two Strategies for Management of Anti-Retroviral Therapy (The SMART Study)
Brief Title: A Study of Anal Cancer Development in HIV Infected People
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 065G; SMART; 10117 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2005-04-06; First posted 2005-04-07 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections; Anus Neoplasms
Keywords: Treatment Experienced; HIV; HPV; Antiretroviral Therapy, Highly Active; Papillomavirus, Human
MeSH Terms: conditions — HIV Infections; Anus Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to compare the development of abnormal cell growth or cancer in the anal region of individuals who are receiving one of two different anti-HIV treatment strategies.

DETAILED DESCRIPTION:
Human papillomavirus (HPV) is a common viral infection among men and women. Individuals with HPV are at risk for anal dysplasia, a condition that may lead to anal cancer. It has been observed that HIV progresses more rapidly in individuals coinfected with HPV and HIV, compared to people with either disease alone. Studies that have investigated the effect of highly active antiretroviral therapy (HAART) on the progression of anal dysplasia have been contradictory and inconclusive. The role of CD4 count and HIV suppression and their contributions to the progression of anal disease needs to be determined. This trial is a substudy of a study of management of antiretroviral therapy (SMART). In the SMART study, patients will participate in one of two strategies: a drug conservation (DC) strategy and a viral suppression (VS) strategy. Participants in the DC group will stop or defer HAART, then receive episodic HAART treatment for the minimum time needed to maintain a CD4 cell count of at least 250 cells/mm3. Participants in the VS group will receive HAART to maintain a viral load as low as possible, regardless of CD4 count. This study will compare the times to development of high-grade anal dysplasia or anal cancer in participants who are currently enrolled in the SMART study.

Patients will participate in this substudy and the main SMART study at the same time. At the baseline visit, participants will undergo an anal swab; some female participants will have a cervical swab as well. Participants will provide a detailed sexual history including sexually transmitted infections, a history of anal-related conditions, and a history of alcohol and recreational drug use. These procedures will be repeated at each annual follow-up visit. Some participants may undergo additional anal cytology and high-resolution anoscopy with biopsy. Participants will be followed until they develop high-grade anal dysplasia or anal cancer or when the SMART study closes, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Coenrollment in the SMART study
* Normal anal cytology result. If baseline anal cytology is abnormal, high-resolution anoscopy must be performed and specimens must be obtained.
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Current or prior history of anal or cervical cancer
* Permanent or irreversible bleeding disorder that would interfere with biopsy of the anal canal

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 560
Dates: Start 2005-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Time to high-grade anal dysplasia or anal cancer

SECONDARY OUTCOMES:
Time to anal cancer
time to low-grade or high-grade anal dysplasia
time to anal HPV infection
time to anal HPV infection with a specific strain, for types 16, 18, or 31
time to cervical HPV infection
time to cervical HPV infection with a specific strain, for types 16, 18, or 31
time to high-grade anal dysplasia
time from low-grade anal dysplasia to normal

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Cohen, MD, MSc, Study Chair — Community Research Initiative of New England
Locations (13):
- United States (13):
  - LA Gay & Lesbian Community Service Ctr., Lamba Med. Group CRS, Los Angeles, California
  - Castro-Mission Health Ctr. CRS, San Francisco, California
  - Univ. of Colorado Health Science Ctr. CRS, Denver, Colorado
  - Eastside Family Health Ctr. CRS, Denver, Colorado
  - Washington DC VAMC, Washington Regional AIDS Program, Infectious Diseases CRS, Washington D.C., District of Columbia
  - Univ. of Florida, Div. of Infectious Diseases CRS, Jacksonville, Florida
  - CRI-Boston CRS, Boston, Massachusetts
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Harlem Hospital Ctr./Columbia University CRS (Gordin CTU), New York, New York
  - Kaiser Immune Deficiency Clinic of Portland CRS, Portland, Oregon
  - Oregon Health & Sciences Univ. Internal Medicine (L-475) CRS, Portland, Oregon
  - Temple Univ. School of Medicine CRS, Philadelphia, Pennsylvania
  - Houston AIDS Research Team CRS, Houston, Texas

REFERENCES:
- [Background] Panther LA, Schlecht HP, Dezube BJ. Spectrum of human papillomavirus-related dysplasia and carcinoma of the anus in HIV-infected patients. AIDS Read. 2005 Feb;15(2):79-82, 85-6, 88, 91. PMID 15712398
- [Background] Heard I, Palefsky JM, Kazatchkine MD. The impact of HIV antiviral therapy on human papillomavirus (HPV) infections and HPV-related diseases. Antivir Ther. 2004 Feb;9(1):13-22. PMID 15040532
- [Background] Piketty C, Darragh TM, Da Costa M, Bruneval P, Heard I, Kazatchkine MD, Palefsky JM. High prevalence of anal human papillomavirus infection and anal cancer precursors among HIV-infected persons in the absence of anal intercourse. Ann Intern Med. 2003 Mar 18;138(6):453-9. doi: 10.7326/0003-4819-138-6-200303180-00008. PMID 12639077
- [Background] Manzione CR, Nadal SR, Calore EE. [Human papillomavirus oncogenicity and grade of anal intraepithelial neoplasia in HIV positive patients]. Rev Assoc Med Bras (1992). 2004 Jul-Sep;50(3):282-5. doi: 10.1590/s0104-42302004000300035. Epub 2004 Oct 21. Portuguese. PMID 15499480
- See also: Click here for more information on CPCRA 065 — http://clinicaltrials.gov/ct/show/NCT00027352